CLINICAL TRIAL: NCT00984971
Title: A Two-site, Phase 1, Partially-blinded, Placebo-controlled Safety, Acceptability and Pharmacokinetic Trial of Topical, Vaginally-formulated Tenofovir 1% Gel Applied Rectally Compared With Oral 300 mg Tenofovir Disoproxil Fumarate in HIV-1 Seronegative Adults
Brief Title: Rectal Microbicide Safety and Acceptability Trial of Topically Applied Tenofovir Compared With Oral Tablet
Acronym: RMP02-MTN006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Microbicide Trials Network (Network)
Responsible Party: Peter A. Anton, MD, UCLA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DAIDS ID 10769; RMP02-MTN006
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: HIV Prevention; HIV Infections
Keywords: Microbicides; Tenofovir; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tenofovir (Experimental)
  Interventions: Drug: Tenofovir
- HEC Placebo (Placebo Comparator)
  Interventions: Drug: HEC Placebo
- Open label tenofovir tablet (Other)
  Interventions: Drug: Open label tenofovir tablet

INTERVENTIONS:
Drug: Tenofovir — Topical gel applied rectally
  Arms: Tenofovir
Drug: HEC Placebo — Placebo gel applied rectally
  Arms: HEC Placebo
Drug: Open label tenofovir tablet — All participants will undergo an open label tenofovir tablet single dose administration (i.e. Tenofovir Disoproxil Fumarate 300 mg, aka Viread®)
  Arms: Open label tenofovir tablet

SUMMARY:
To date, the majority of microbicide research has focused on the assessment of the safety and effectiveness of vaginal microbicides used for the prevention of HIV transmission via the vaginal compartment. Receptive anal intercourse (RAI) is common among men who have sex with men (MSM), and there is increasing evidence that heterosexual women in the developed and developing world also practice anal sex. It can, therefore, be anticipated that once vaginal microbicides are licensed, they will be used in both the vaginal and rectal compartments. As a consequence, there is a need to evaluate both the rectal and vaginal safety profile of candidate microbicides. Therefore, the primary objective of this study is to evaluate the systemic safety of 1% vaginally formulated tenofovir gel applied rectally. In addition, this study will evaluate the immunotoxicity of the gel and evaluate its acceptability; it will also use the oral tenofovir disoproxil fumarate tablets (TDF), rectally-applied tenofovir gel,and a placebo gel to compare their systemic and compartmental pharmacokinetic (pK) profiles.

This study was designed to address the following hypotheses:

* Vaginally-formulated tenofovir 1% topical gel when applied rectally will be safe using a combination of clinical and laboratory markers including assays specifically designed to measure mucosal toxicity
* Tenofovir will be detectable at different concentrations in the various anatomic compartments sampled for pharmacokinetics following single and 7-day topical exposures
* Exposure to tenofovir 1% gel will demonstrate prevention of ex vivo HIV-1 challenge using in vivo drug-exposed tissue as compared to baseline tissue samples
* Orally delivered, single dose, 300 mg tenofovir disoproxil fumarate tablets will have similar safety profiles using routine blood safety indices as have been established in other trials and will show no mucosal safety concerns
* The oral dose will have different multi-compartment concentration kinetics than the topical tenofovir and will also demonstrate preliminary (ex vivo) prevention using the explant infectivity assay
* Vaginally formulated tenofovir 1% topical gel applied rectally will be acceptable to participants, as indicated by a score in the upper one third of the 10-point Likert scale on intentionality to use in the product in the future

ELIGIBILITY:
Inclusion Criteria

1. ≥ Age of 18 at screening
2. Willing and able to provide written informed consent for screening and enrollment
3. HIV-1 uninfected at screening according to the standard DAIDS algorithm in Appendix II
4. Willing and able to communicate in English
5. Willing and able to provide adequate locator information, as defined in site standard operating procedures (SOP)
6. Availability to return for all study visits, barring unforeseen circumstances
7. Per participant report at screening, a history of consensual RAI at least once in the prior year
8. Willing to abstain from insertion of anything rectally including sex toys, other than the study gel during the active phases of the study and for 5 days following biopsy collection
9. Willing to abstain from sexual intercourse (rectal and vaginal) during the active phases of the study and for 5 days following biopsy collection
10. Must agree to use study provided condoms for the duration of the study for vaginal and insertive anal intercourse
11. Must be in general good health
12. Must agree not to participate in other drug trials

    In addition to the criteria listed above, female participants must meet the following criteria:
13. Post-menopausal or using (or willing to use) an acceptable form of contraception (e.g., barrier method, IUD, hormonal contraception, surgical sterilization, or vasectomization of male partner). If the female participant has female partners only, the method of contraception will be noted as a barrier method in the study documentation.

Exclusion Criteria

1. Abnormalities of the colorectal mucosa, or significant colorectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids)
2. At screening, clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines or urinary tract infection (UTI). Infections requiring treatment include symptomatic bacterial vaginosis, symptomatic vaginal candidiasis, other vaginitis, trichomoniasis, Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, pelvic inflammatory disease, genital sores or ulcers, cervicitis, or symptomatic genital warts requiring treatment. Note that HSV-2 seropositive with no active lesions is allowed, since treatment is not required.

   Note: Allow one re-screening after documented treatment (30 days) in cases of GC/CT identified at screening
3. At screening:

   1. Positive for hepatitis B surface antigen
   2. Hemoglobin < 10.0 g/dL
   3. Platelet count < 100,000/mm3
   4. White blood cell count less than 2,000 cells/mm3 or > than 15,000 cells/mm3
   5. Calculated creatinine clearance less than 80 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min (140- age in years) x (weight in kg) x (0.85 for females)/72 x (serum creatinine in mg/dL)
   6. Serum creatinine > 1.3× the site laboratory upper limit of normal (ULN)
   7. ALT and/or AST > 2.5× the site laboratory ULN
   8. +1 glucose or +1 protein on urinalysis (UA)
   9. History of bleeding problems (i.e. INR > 1.5× the site laboratory ULN or PTT > 1.25× the site laboratory ULN)
4. History of significant gastrointestinal bleeding in the opinion of the investigator
5. Allergy to methylparaben, propylparaben, sorbic acid
6. By participant report at enrollment, history of excessive daily alcohol use (as defined by the CDC as heavy drinking consisting of an average consumption of more than 2 drinks per day for men, and more than 1 drink per day for women), frequent binge drinking or illicit drug use that includes any injection drugs, methamphetamines (crystal meth), heroin, or cocaine including crack cocaine, within the past 12 months
7. Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation:

   1. Heparin, including Lovenox®
   2. Warfarin
   3. Plavix® (clopidogrel bisulfate)]
   4. Rectally administered medications (including over-the-counter products)
   5. Aspirin
   6. NSAIDS
   7. Acyclovir
   8. Valacyclovir
   9. TDF
   10. Any other drugs that are associated with increased likelihood of bleeding following mucosal biopsy
8. By participant report at screening, use of systemic immunomodulatory medications, rectally administered medications, rectally administered products (including condoms) containing N-9, or any investigational products within the 4 weeks prior to the Enrollment/Baseline Evaluation Visit
9. History of recurrent urticaria
10. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.

    In addition to the criteria listed above, female participants will be excluded if they meet any of the following criteria:
11. Pregnant at Enrollment/Baseline Evaluation Visit
12. Breastfeeding or intent to breastfeed during duration of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Grade 2 or higher clinical and laboratory adverse events as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0,Dec 2004 and Addenda 1 and 3 to this table. | Every study visit

SECONDARY OUTCOMES:
Immunotoxicity, Pharmacokinetics, and Acceptability | Immunotoxicity and pharmacokinetics: every study visit; acceptability: baseline and end of study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Center for HIV Prevention Research, Los Angeles, California
  - University of Pittsburgh Clinical Research Unit, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Richardson-Harman N, Hendrix CW, Bumpus NN, Mauck C, Cranston RD, Yang K, Elliott J, Tanner K, McGowan I, Kashuba A, Anton PA. Correlation between compartmental tenofovir concentrations and an ex vivo rectal biopsy model of tissue infectibility in the RMP-02/MTN-006 phase 1 study. PLoS One. 2014 Oct 28;9(10):e111507. doi: 10.1371/journal.pone.0111507. eCollection 2014. PMID 25350130
- [Derived] Yang KH, Hendrix C, Bumpus N, Elliott J, Tanner K, Mauck C, Cranston R, McGowan I, Richardson-Harman N, Anton PA, Kashuba AD. A multi-compartment single and multiple dose pharmacokinetic comparison of rectally applied tenofovir 1% gel and oral tenofovir disoproxil fumarate. PLoS One. 2014 Oct 28;9(10):e106196. doi: 10.1371/journal.pone.0106196. eCollection 2014. PMID 25350119
- [Derived] Anton PA, Cranston RD, Kashuba A, Hendrix CW, Bumpus NN, Richardson-Harman N, Elliott J, Janocko L, Khanukhova E, Dennis R, Cumberland WG, Ju C, Carballo-Dieguez A, Mauck C, McGowan I. RMP-02/MTN-006: A phase 1 rectal safety, acceptability, pharmacokinetic, and pharmacodynamic study of tenofovir 1% gel compared with oral tenofovir disoproxil fumarate. AIDS Res Hum Retroviruses. 2012 Nov;28(11):1412-21. doi: 10.1089/aid.2012.0262. Epub 2012 Oct 9. PMID 22943559
- [Derived] Richardson-Harman N, Mauck C, McGowan I, Anton P. Dose-response relationship between tissue concentrations of UC781 and explant infectibility with HIV type 1 in the RMP-01 rectal safety study. AIDS Res Hum Retroviruses. 2012 Nov;28(11):1422-33. doi: 10.1089/AID.2012.0073. Epub 2012 Sep 20. PMID 22900504